CLINICAL TRIAL: NCT04355624
Title: Characterization of Kidney Involvement in COVID-19 Disease: a French Multi-center Prospective Observational Study
Brief Title: Kidney Involvement in COVID-19 Disease (COVKID)
Acronym: COVKID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20reamedcovid02
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: COVID; Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and urine. Renal tissue only from post-portem kidney biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU patients: COVID-19 patients admitted in Intensive Care Units
- Non ICU patients: COVID-19 patients admitted in conventional units

SUMMARY:
Novel coronavirus disease (COVID-19) is a newly discovered contagious disease caused by SARS-CoV-2 virus, primarily manifesting as an acute respiratory illness with pneumonia, but can affect multiple organs such as kidney, heart, digestive tract, blood and nervous system. In previous reports of SARS and MERS-CoV infections, acute kidney injury was described in 5 to 15% of patients and was associated with a high mortality rate (60-90%). Recent reports showed renal abnormalities in COVID-9 infected patients. A recent Chinese study also reported that acute kidney injury was an independent risk factor for mortality. However, the exact mechanism of kidney involvement remains unclear: sepsis-related cytokine storm or direct cellular injury from the virus. Also, kidney involvement has not yet been well characterized: heavy albuminuria, hematuria or interstitial nephropathy alone.

A recent study identified viral RNA in kidney tissue and another study succeeded isolating SARS-CoV-2 from the urine sample of an infected patient. These data suggest that the kidney might be a target of this novel coronarivus.

The sponsor suggests characterizing kidney involvement in SARS-CoV-2 infection.

Study objectives are:

* To give an accurate characterization of kidney involvement in COVID-19
* To investigate the physiopathologic mechanism of kidney involvement in SARS-CoV-2 infection
* To identify risk factors for kidney involvement in in SARS-CoV-2 infection
* To evaluate the impact of kidney involvement in in SARS-CoV-2 infection
* To assess the long-term health effect of kidney injury on survivors of in SARS-CoV-2 infection

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 disease
* Age > 18 years-old

Exclusion Criteria:

* Age < 18 years-old
* Pregnancy
* Patient with tutor- or curatorship or in prison
* Patients who had undergone renal replacement therapy (RRT) before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 disease
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Kidney involvement in COVID-19 disease | until 3 months after discharge or death
  Rate of kidney involvement in COVID-19 disease characterized by clinical and biological data

SECONDARY OUTCOMES:
Physiopathologic mechanism of kidney involvement in SARS-CoV-2 infection | until 3 months after discharge or death
  biological data and histopathological data if available
To identify risk factors for kidney involvement in in SARS-CoV-2 infection | until 3 months after discharge or death
  Rate of death
To evaluate the impact of kidney involvement in SARS-CoV-2 infection | until 3 months after discharge or death
  Legnth of hopital stay
To assess the long-term health effect of kidney injury on survivors of SARS-CoV-2 infection in case of AKI KDIGO 2 or 3 | until 3 months after discharge
  Recovery of Kidney fonction

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre hospitalier d'Antibes Juan les pins, Antibes
  - Centre hospitalier de Cannes, Cannes
  - Centre hospitalier de Grasse, Grasse
  - CHU de Nice, Nice

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established